CLINICAL TRIAL: NCT06760910
Title: Efficacy of Transcranial Direct Current Stimulation in the Amblyopia Treatment of Older Adolescents: A Cohort Study
Brief Title: Clinical Treatment of Transcranial Direct Current Stimulation in Older Adolescents With Amblyopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Principal Investigator, Yatu Guo, Principal Investigator, Tianjin Eye Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YK2023001
Record Dates: First submitted 2024-03-25; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Amblyopia
Keywords: Amblyopia; transcranial direct current stimulation(tDCs); adolescent; treatment
MeSH Terms: conditions — Amblyopia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS Group (Active Comparator): Participants will receive anodal transcranial direct current stimulation (tDCS) with electrodes placed over the occipital cortex, chosen due to its critical role in processing visual information and its potential responsiveness to neuromodulation in amblyopia treatment. The stimulation will be set at 0.1 mA for 20 minutes per session, twice a week, over 6 months
  Interventions: Procedure: tDCS Stimulation; Device: Anodal tDCS
- Sham Stimulation Group (Sham Comparator): Participants will receive sham tDCS with electrodes similarly placed over the occipital cortex. The stimulation will be set at 0 mA for 20 minutes per session, twice a week, over 6 months
  Interventions: Procedure: tDCS Stimulation; Device: Sham tDCS

INTERVENTIONS:
Procedure: tDCS Stimulation — Anode tDCS or sham stimulation for amblyopia of Adolescents
Device: Anodal tDCS — Anodal tDCS
  Arms: Anodal tDCS Group
Device: Sham tDCS — Sham tDCS
  Arms: Sham Stimulation Group

SUMMARY:
As a neurodevelopmental visual disorder, amblyopia, especially monocular form-deprivation amblyopia, can lead to severe visual developmental impairments. Due to reduced neural plasticity in the visual cortex after the critical period of visual development, older children and adults with amblyopia show poor responses to conventional treatments, lacking effective therapeutic options. Recent basic and clinical research has shown that transcranial direct current stimulation can effectively treat adult amblyopia by altering cortical excitability, enhancing synaptic plasticity, and affecting the excitatory/inhibitory balance in the cortex to reboot adult visual cortex plasticity. This proposed study aims to conduct a large-scale prospective randomized controlled trial to objectively assess the efficacy and safety of transcranial direct current stimulation in treating amblyopia in older adolescents and adults. By comparing changes in best-corrected visual acuity, visual evoked potentials(VEPs), contrast sensitivity, and functional connectivity between the visual cortex and other cortical areas using fMRI, the study seeks to provide robust clinical evidence, clarify the treatment effects of transcranial direct current stimulation in adult amblyopia, elucidate potential mechanisms of enhancing adult visual cortex plasticity with transcranial direct current stimulation, and potentially offer a safe and effective treatment modality for adult amblyopia.

DETAILED DESCRIPTION:
1. A prospective cohort study designed to evaluate the effectiveness of transcranial direct current stimulation (tDCS) in improving visual outcomes in older adolescents with amblyopia. Anodal tDCS Group: Participants will receive anodal transcranial direct current stimulation (tDCS) with electrodes placed over the occipital cortex, chosen due to its critical role in processing visual information and its potential responsiveness to neuromodulation in amblyopia treatment. The stimulation will be set at 0.1 mA for 20 minutes per session, twice a week, over 6 months; Sham Stimulation Group: Participants will receive sham tDCS with electrodes similarly placed over the occipital cortex. The stimulation will be set at 0 mA for 20 minutes per session, twice a week, over 6 months.
2. The impact of transcranial direct current stimulation on adult visual cortex plasticity and cortical functional assessment. Before and after transcranial direct current stimulation, resting-state and task-based functional magnetic resonance imaging (fMRI) are used to assess the functional activity between the visual cortex and other cortical regions. This evaluation aims to identify changes in adult visual cortex plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Children and their legal guardians have obtained consent in writing.
* Participants aged 10-30, of any gender.
* Participants must meet the diagnostic criteria for amblyopia: unilateral amblyopia with a difference of two lines or more in visual acuity between the eyes, or bilateral amblyopia with best-corrected visual acuity worse than 20/30 (or worse than 0.2 logMAR). The visual acuity charts to be used are LEA SYMBOLS® (Good-Lite Co., Elgin, IL) or HOTV visual acuity chart.

Exclusion Criteria:

* Participants who may have eye diseases affecting vision or refractive errors (such as cataracts, crystalline lens damage, glaucoma, macular degeneration, corneal disorders, retinitis pigmentosa, retinal detachment, severe vitreous opacities, etc
* History of eye trauma or intraocular surgery
* Inability to cooperate with examinations
* Presence of concomitant systemic diseases (such as epilepsy)
* Participation in any other experimental treatment within the past 3 months
* Other situations deemed unsuitable by the investigator.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in Best Corrected Visual Acuity (BCVA) | 24 weeks
  quantified by the number of lines gained on a standard visual acuity chart(HOTV chart). This measure will be assessed at baseline, 3 months, and 6 months post-intervention. A line gain is defined as the ability to correctly read an additional row of optotypes compared to baseline measurements. The improvement will be evaluated separately for each eye and averaged to assess overall treatment efficacy.

SECONDARY OUTCOMES:
Changes in Visual Evoked Potential (VEP) | 24 weeks
  changes in Visual Evoked Potential (VEP) metrics, specifically amplitude and latency, at 15 minutes and 1-degree visual angle stimulations. These measures will be used to assess the functional responsiveness of the visual pathways and cortical processing efficiency. Baseline, 3-month, and 6-month assessments will provide comparative data to evaluate the neurophysiological effects of the intervention.
Improvements in contrast sensitivity at different spatial frequencies | 24 weeks
  Contrast sensitivity will be evaluated using a contrast sensitivity test with CSV-1000E(Vector vision, US), which measures the ability to detect differences in luminance across varying spatial frequencies (low 3 c/d, medium 6c/d、12 c/d, and high 18 c/d). Assessments will be conducted at baseline, 3 months, and 6 months post-intervention. The degree of improvement will be compared across groups to determine the impact of tDCS on visual function beyond acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No